CLINICAL TRIAL: NCT06254235
Title: Bioequivalence Study of Octreotide Acetate Microsphere Injection in Human
Brief Title: Bioequivalence Study of Two Octreotide Microsphere Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QL-YXZ2-006
Record Dates: First submitted 2024-01-22; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental)
  Interventions: Drug: The test octreotide microsphere
- Reference (Active Comparator)
  Interventions: Drug: The reference octreotide microsphere

INTERVENTIONS:
Drug: The test octreotide microsphere — A single intramuscular dose of the test octreotide microsphere 30mg,
  Arms: Test
Drug: The reference octreotide microsphere — A single intramuscular dose of the reference octreotide microsphere 30mg
  Arms: Reference

SUMMARY:
The goal of this clinical trial is to evaluate the pharmacokinetic characteristics of two octreotide microsphere formulations in healthy Chinese volunteers.

Participants will receive single-dose of either test or reference octreotide microsphere formulations.

Researchers will compare pharmacokinetic characteristics of the two formulations to see if they are bioequivalent.

ELIGIBILITY:
Inclusion Criteria:

* BMI 19-28 kg/m^2, and with weight ≥ 50 kg for male, or ≥ 45 kg for female
* In good physical condition (without any history of disease or clinically relevantly abnormal vital sign or examination
* Agreed to use adequate contraception and did not plan for pregnancy from screening period throughout 6 months after study completion
* Fully understood and voluntarily signed the informed consent form
* With high compliance

Exclusion Criteria:

* With allergic disease or allergic to any component of the study drugs or more than two kinds of other drug, food, or beverage
* Positive for human immunodeficiency virus, hepatitis B, C, or syphilis test
* With gastrointestinal disease
* Had drug addiction within 5 years or used narcotics within 6 months before screening or positive in drug of abuse test
* With alcohol consumption > 2 units/d within 6 months before screening
* With cigarette consumption > 5/d within 3 months before screening
* Donated or lost blood > 400 mL within 3 months before screening
* Hospitalized or received surgery within 3 months before screening
* Received study drug of other clinical trial within 3 months before screening
* Received prescription drug within 14d before dosing
* Received over-the-counter drug or herb within 48h before dosing
* Consumed grape fruit juice, or other food or beverage containing caffeine or xanthine within 72h before dosing
* Consumed alcohol within 48h before dosing or positive for breath alcohol test
* Cannot consume standard meal
* Intolerable to venipuncture
* Cannot receive intramuscular injection in the glute
* With vitamin B12 deficiency
* Had acute minor disease (common cold, diarrhea, etc.) from screening to dosing
* For pregnancy-capable female, breastfeeding or positive for pregnancy test at screening, or had unprotected sexual contact within 2 weeks before dosing
* Other reason judged by investigators

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
AUC0-28d | Day 0-28
  The area under the concentration-time curve from dosing to Day 28
AUC28-56d | Day 28-56
  The area under the concentration-time curve from Day 28 to Day 56
AUC0-t | Day 0-82
  The area under the concentration-time curve from dosing to the last quantifiable time-point
AUC0-∞ | Day 0-82
  The area under the concentration-time curve extrapolated to infinity
Cmax | Day 0-82
  The maximum drug concentration

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China